CLINICAL TRIAL: NCT02819960
Title: Prevention of Irinotecan Induced Diarrhea by Probiotics: A Phase III Study
Brief Title: Prevention of Irinotecan Induced Diarrhea by Probiotics
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: S&D Pharma SK s.r.o. (Industry)
Collaborators: National Cancer Institute, Slovakia (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2
Record Dates: First submitted 2016-05-11; First posted 2016-06-30 (Estimated); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: Diarrhea; Cancer
Keywords: probiotics; irinotecan; diarrhea; Lactobacillus rhamnosus; Bifidobacterium animalis; prevention; chemotherapy
MeSH Terms: conditions — Diarrhea; Neoplasms | interventions — maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- active probiotic formula (Active Comparator): Intervention: Probiotic formula Probio-Tec® BG-VCap-6.5 will be administered at a dose of 3x1 cps per day orally for 6 weeks. No premedication or patient monitoring after administration of probiotic formula is required. Probiotic formula may be taken after meals or snacks to reduce stomach upset. Swallow the capsule or in case of problems with swallowing, capsule can be opened, content mixed with small amount of food. Food must not be hot.
  Patients should receive full supportive care during the study, including transfusion of blood and blood products, treatment with antibiotics, anti-emetics, anti-diarrheal agents, analgesics, erythropoetin, or bisphosphonates, when appropriate.
  Interventions: Drug: Probio-Tec® BG-VCap-6.5
- placebo (Placebo Comparator): Intervention: Maltodextrin will be used for placebo group and will be administered at a the same dose as active formula (3x1 cps per day orally for 6 weeks).
  Patients should receive full supportive care during the study, including transfusion of blood and blood products, treatment with antibiotics, anti-emetics, anti-diarrheal agents, analgesics, erythropoetin, or bisphosphonates, when appropriate.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Probio-Tec® BG-VCap-6.5 — Each capsule contents: 2 lyophilized probiotic strains, total amount of minimum 2,7x10 9 CFU/cps, ratio LGG®: BB-12® = 50% : 50% (Culture percentages are based on cell concentration and are approximate) Lactobacillus rhamnosus GG® (ATCC 53103) Bifidobacterium animalis subsp. lactis BB-12® (DSM 15954) Additives: maltodextrin, microcrystalline cellulose, silicium dioxide, magnesium stearate
  Other Names: PROBIO-FIX INUM®
  Arms: active probiotic formula
Drug: Placebo — Maltodextrin
  Other Names: Maltodextrin
  Arms: placebo

SUMMARY:
Diarrhea is a relatively common complication in patients with cancer. At its inception, several mechanisms participated; malabsorption on the basis of mucositis induced by chemotherapy, dysbiosis induced by broad-spectrum antibiotics and predisposition to infectious diarrhea in immunocompromised patients. Some cytostatics and their metabolites can also induce diarrhea directly due to effect on the intestinal mucosa.

Use of probiotics in prevention and treatment of diarrhea relies on both the theoretical assumptions and the results of several clinical trials. Lactic acid bacteria involved in the treatment of dysbiosis, compete for substrate with pathogenic bacteria, produce bacterio-cins, increase transepithelial resistance. Their enzymatic activity affects activation or deactivation of metabolites which cause diarrhea. Production of short chain fatty acids, which are important for the maintenance of intestinal mucosal cells also contributes to their antidiarrhoeal effect.

This randomized, double-blind, placebo controlled, multicentre trial was designed to evaluate potential of probiotics to prevent grade 3-4 diarrhea in patients treated by irinotecan based chemotherapy during first 6 weeks of irinotecan based chemotherapy

DETAILED DESCRIPTION:
In preventing antibiotic-induced diarrhea in double blind placebo controlled clinical trials it was found protective effect of probiotics containing S. boulardii and Enterococcus faecium. Also in preventing infectious diseases associated with Clostridium difficile, administration of probiotics resulted in a significant decrease in disease recurrence. Duration of rotavirus diarrhea, in children and in immunocompromised HIV-positive patients was significantly shortened after administration of strains of Lactobacilli and S. boulardii respectively.

Meta-analysis of 9 randomized, placebo-controlled trials showed significant reduction in the incidence of antibiotic associated diarrhea in children. Another meta-analysis in which 23 studies were included showed significant reduction in risk of infectious diarrhea. Most of these studies was carried out with the probiotic strain Lactobacillus rhamnosus GG®.

The incidence of diarrhea during treatment of acute leukemia is between 15 to 80%. Severe diarrhea level 3 to 4 is present in 8-20% and is much more common during the induction phase of chemotherapy. In phase II study performed in NCI Slovakia preventive administration of Enterococcus faecium probiotic strain M-74 with selenium was associated with low incidence (14%) and severity (all grade 1) diarrhea, despite the fact that half of the patients received induction therapy. The investigators noted safety of probiotic strain during 370 days of severe neutropenia Gr 3-4.

The incidence of irinotecan induced diarrhea varies between 60-90%, by which the incidence of severe diarrhea is 20-40%. In phase II studies, its incidence was 17% in NCI Slovakia, but irinotecan dose was reduced by 25% in all patients. Diarrhea is an important factor in morbidity and mortality during irinotecan based chemotherapy. Predisposing factors are age over 65 years, ECOG (Eastern Cooperative Oncology Group) PS (Performance status) of 1 and previous abdominopelvic radiation. One of irinotecan metabolites, SN-38 (7-ethyl-10 hydroxycamptothecin), which is glucuronidated in the liver and subsequently expelled into intestine is main cause of diarrhea. Due to the bacterial enzyme beta-D-glucuronidase it is deconjugated in intestinal lumen again. This form causes direct damage to intestinal mucosa associated with malabsorption of water, electrolytes and development of diarrhea.

Reduction of activity of intestinal beta-D-glucuronidase using broad-spectrum antibiotics and/or beta-D-glucuronidase inhibitors is one of the ways to avoid irinotecan induced diarrhea. It is also possible to modulate metabolism of irinotecan using cyclosporine and phenobarbital to reduce biliary excretion of SN-38 and induction of glucuronidation. Promising results were shown using activated charcoal, which has resulted in the absorption of SN-38. Also other methods were tested: oral alkalization, thalidomide, amifostine, but without success. These procedures have been studied only in phase II trials. It is known that some probiotic bacteria, reduce activity of intestinal beta-D-glucuronidase and therefore these bacteria could be applied in the prevention of diarrhea in patients treated by irinotecan based therapy.

Results of phase III study, that was prematurely terminated due to poor accrual showed benefit of Colon Dophilus on irinotecan induced gastrointestinal toxicity. In this trial, 46 patients with colorectal cancer starting a new line of irinotecan based therapy were enrolled. 5-fluorouracil/capecitabine along with irinotecan was administered to 26 (56.5%) patients and 22 (47.8%) patients received biological therapy as well. Patients were randomized 1:1 to probiotic (PRO) or placebo arm (PLA). Probiotic formula Colon Dophilus, was administered at a dose of 10x109 CFU (colony forming unit) of bacteria tid, orally for 12 weeks of chemotherapy. Primary endpoint was incidence of grade 3/4 diarrhea. 23 patients were randomized to PRO and 23 patients to PLA. Administration of probiotics compared to placebo led to a reduction in the incidence of severe diarrhea of grade 3 or 4 (0% for PRO vs. 17.4% for PLA, p = 0.11), as well as reduction of the overall incidence of diarrhea (39.1% for PRO vs. 60.9% for PLA, p = 0.24) and incidence of enterocolitis (0% for PRO vs. 8.7% for PLA). Patients on PRO used less loperamide compared to PLA (mean duration of loperamide use: 4.5 days for PRO vs. 10.4 days for PLA, p = 0.45; mean number of loperamide tablets: 5.9 for PRO vs. 37.7 for PLA, p = 0.49). There was no infection caused by probiotic strains recorded.

Two recent studies in murine model showed, that bacteria in the gut enhance the body's immune response to cancer, mobilizing immune cells to kill cancer cells, not just in the gut but throughout the body as well. The researchers also found that the bacteria affect the efficacy of three different cancer treatments.

Given their low toxicity, good tolerability, probiotics may be an important part of supportive therapy and moreover they can enhance efficacy of anticancer therapy. The objective of this phase III. trial is to determine effectiveness of the probiotic formula Probio-Tec® BG-VCap-6.5 in the prophylaxis of irinotecan induced diarrhea due to reduction intestinal beta-D-glucuronidase activity and further biochemical and physiological actions of specific strains Bifidobacterium animalis subsp. lactis BB-12® and Lactobacillus rhamnosus GG®, LGG® that are active substances of used food supplement - PROBIO-FIX INUM®. Both of strains are well-documented. LGG® has been studied in more over 800 scientific publications. Studies have found that LGG® supports immunity, enhances antibody formation during viral infection, and decreases incidence of gastrointestinal infections, antibiotic associated diarrhoea, and respiratory infections. In addition to its well-researched health benefits, the safety of LGG® has been more widely studied than any other probiotic bacterium. It has a safe history of use in foods and is extensively documented in more over 200 clinical studies.

The large number of clinical studies and scientific publications indicate that the BB-12® probiotic strain - alone or in combination with other of probiotic strains (e.g. LGG®) - may have beneficial effects regarding the gastrointestinal and immune areas. BB-12® is considered to be best studied probiotic bifidobacteria, described in more than 360 scientific studies.

ELIGIBILITY:
Inclusion Criteria:

* signed written informed consent
* age > 18 years
* histologically proven colorectal cancer patients starting new line of chemotherapy based on irinotecan
* ECOG PS 0 - 1 at study entry
* life expectancy more than 3 months
* absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule;

Exclusion Criteria:

* impossibility to take oral medication
* active infection treated by antibiotic therapy
* ileostoma
* hypersensitivity to study drug
* any concurrent malignancy other than non-melanoma skin cancer, no other cancer in past 5 years.
* serious concomitant systemic disorders or diseases incompatible with the study (at the discretion of investigator )

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 233 (Actual)
Dates: Start 2016-03; Primary Completion 2022-08 (Actual); Study Completion 2022-11 (Actual)

PRIMARY OUTCOMES:
Prevention of grade 3-4 diarrhea induced by irinotecan based chemotherapy | first 6 weeks of irinotecan based chemotherapy
  To determine the efficacy (as measured by prevention of grade 3/4 diarrhea) of probiotic formula Probio-Tec® BG-VCap-6.5 given orally to patients with colorectal cancer starting new line of irinotecan based chemotherapy. Response will be defined as prevention of grade 3/4 diarrhea according to definition of NCI CTC version 4.0

SECONDARY OUTCOMES:
Progression-free survival | 1 year
  Progression-free survival period will be evaluated according to standard protocol.
Prevention of any grade of diarrhea | 6 weeks
  To determine the efficacy (as measured by prevention of grade 1/2 diarrhea) of probiotic formula Probio-Tec® BG-VCap-6.5 given orally to patients with colorectal cancer during first 6 weeks of irinotecan based chemotherapy. Response will be defined as prevention of grade 1/2 diarrhea according to definition of NCI CTC version 4.0
Prevention of other gastrointestinal symptoms | 6 weeks
  To determine the efficacy (as measured by prevention of enterocolitis) of probiotic formula Probio-Tec® BG-VCap-6.5 given orally to patients with colorectal cancer starting new line of irinotecan based chemotherapy. Response will be defined as prevention of enterocolitis during first 6 weeks of irinotecan based chemotherapy according to definition of NCI CTC version 4.0.
Incidence of treatment-emergent adverse events [Safety and Toxicity] | 6 weeks
  Safety and toxicity will be evaluated according to NCI Common Terminology Criteria for Adverse Events Version 4.0 (CTCAE) (see Appendix D; http://www.fda.gov/cder/cancer/toxicityframe.htm).

CONTACTS AND LOCATIONS:
Overall Officials: Michal Mego, MD, Principal Investigator — National Cancer Institute Bratislava; Lubos Drgona, MD, Principal Investigator — National Cancer Institute Bratislava
Locations (1):
- National Cancer Institute, Bratislava, Slovakia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Batt RM, Rutgers HC, Sancak AA. Enteric bacteria: friend or foe? J Small Anim Pract. 1996 Jun;37(6):261-7. doi: 10.1111/j.1748-5827.1996.tb02376.x. PMID 8805096
- [Background] Born P, Lersch C, Zimmerhackl B, Classen M. [The Saccharomyces boulardii therapy of HIV-associated diarrhea]. Dtsch Med Wochenschr. 1993 May 21;118(20):765. No abstract available. German. PMID 8500427
- [Background] Camera A, Andretta C, Villa MR, Volpicelli M, Picardi M, Rossi M, Rinaldi CR, Della Cioppa P, Ciancia R, Selleri C, Rotoli B. Intestinal toxicity during induction chemotherapy with cytarabine-based regimens in adult acute myeloid leukemia. Hematol J. 2003;4(5):346-50. doi: 10.1038/sj.thj.6200304. PMID 14502260
- [Background] D'Souza AL, Rajkumar C, Cooke J, Bulpitt CJ. Probiotics in prevention of antibiotic associated diarrhoea: meta-analysis. BMJ. 2002 Jun 8;324(7350):1361. doi: 10.1136/bmj.324.7350.1361. PMID 12052801
- [Background] Ebringer L, Ferencik M, Lahitova N, Kacani L, Michalkova D. Anti-mutagenic and immuno-stimulatory properties of lactic acid bacteria. World J Microbiol Biotechnol. 1995 May;11(3):294-8. doi: 10.1007/BF00367102. PMID 24414651
- [Background] Ferencik M, Ebringer L, Mikes Z, Jahnova E, Ciznar I. [Successful modification of human intestinal microflora with oral administration of lactic acid bacteria]. Bratisl Lek Listy. 1999 May;100(5):238-45. Slovak. PMID 10500327
- [Background] Fuller R. Probiotics in man and animals. J Appl Bacteriol. 1989 May;66(5):365-78. PMID 2666378
- [Background] Goldin BR. Intestinal microflora: metabolism of drugs and carcinogens. Ann Med. 1990 Feb;22(1):43-8. doi: 10.3109/07853899009147240. PMID 1970483
- [Background] Iida N, Dzutsev A, Stewart CA, Smith L, Bouladoux N, Weingarten RA, Molina DA, Salcedo R, Back T, Cramer S, Dai RM, Kiu H, Cardone M, Naik S, Patri AK, Wang E, Marincola FM, Frank KM, Belkaid Y, Trinchieri G, Goldszmid RS. Commensal bacteria control cancer response to therapy by modulating the tumor microenvironment. Science. 2013 Nov 22;342(6161):967-70. doi: 10.1126/science.1240527. PMID 24264989
- [Background] Isolauri E, Juntunen M, Rautanen T, Sillanaukee P, Koivula T. A human Lactobacillus strain (Lactobacillus casei sp strain GG) promotes recovery from acute diarrhea in children. Pediatrics. 1991 Jul;88(1):90-7. PMID 1905394
- [Background] McFarland LV, Surawicz CM, Greenberg RN, Fekety R, Elmer GW, Moyer KA, Melcher SA, Bowen KE, Cox JL, Noorani Z, et al. A randomized placebo-controlled trial of Saccharomyces boulardii in combination with standard antibiotics for Clostridium difficile disease. JAMA. 1994 Jun 22-29;271(24):1913-8. PMID 8201735
- [Background] McFarland LV, Surawicz CM, Greenberg RN, Elmer GW, Moyer KA, Melcher SA, Bowen KE, Cox JL. Prevention of beta-lactam-associated diarrhea by Saccharomyces boulardii compared with placebo. Am J Gastroenterol. 1995 Mar;90(3):439-48. PMID 7872284
- [Background] Mego M, Ebringer L, Drgona L, Mardiak J, Trupl J, Greksak R, Nemova I, Oravcova E, Zajac V, Koza I. Prevention of febrile neutropenia in cancer patients by probiotic strain Enterococcus faecium M-74. Pilot study phase I. Neoplasma. 2005;52(2):159-64. PMID 15800715
- [Background] Mego M, Koncekova R, Mikuskova E, Drgona L, Ebringer L, Demitrovicova L, Nemova I, Trupl J, Mardiak J, Koza I, Zajac V. Prevention of febrile neutropenia in cancer patients by probiotic strain Enterococcus faecium M-74. Phase II study. Support Care Cancer. 2006 Mar;14(3):285-90. doi: 10.1007/s00520-005-0891-7. Epub 2005 Sep 21. PMID 16175356
- [Background] Mego M, Chovanec J, Vochyanova-Andrezalova I, Konkolovsky P, Mikulova M, Reckova M, Miskovska V, Bystricky B, Beniak J, Medvecova L, Lagin A, Svetlovska D, Spanik S, Zajac V, Mardiak J, Drgona L. Prevention of irinotecan induced diarrhea by probiotics: A randomized double blind, placebo controlled pilot study. Complement Ther Med. 2015 Jun;23(3):356-62. doi: 10.1016/j.ctim.2015.03.008. Epub 2015 Apr 4. PMID 26051570
- [Background] Michael M, Brittain M, Nagai J, Feld R, Hedley D, Oza A, Siu L, Moore MJ. Phase II study of activated charcoal to prevent irinotecan-induced diarrhea. J Clin Oncol. 2004 Nov 1;22(21):4410-7. doi: 10.1200/JCO.2004.11.125. PMID 15514383
- [Background] Mikes A, Ferencik M, Jahnova E, Ebringer L, Ciznar I. Hypocholesterolemic and immunostimulatory effects of orally applied Enterococcus faecium M-74 in man. Folia Microbiol (Praha). 1995;40(6):639-46. doi: 10.1007/BF02818522. PMID 8768254
- [Background] Resta-Lenert S, Barrett KE. Live probiotics protect intestinal epithelial cells from the effects of infection with enteroinvasive Escherichia coli (EIEC). Gut. 2003 Jul;52(7):988-97. doi: 10.1136/gut.52.7.988. PMID 12801956
- [Background] Saint-Marc T, Rossello-Prats L, Touraine JL. [Efficacy of Saccharomyces boulardii in the treatment of diarrhea in AIDS]. Ann Med Interne (Paris). 1991;142(1):64-5. No abstract available. French. PMID 2048880
- [Background] Sakata Y, Suzuki H, Kamataki T. [Preventive effect of TJ-14, a kampo (Chinese herb) medicine, on diarrhea induced by irinotecan hydrochloride (CPT-11)]. Gan To Kagaku Ryoho. 1994 Jul;21(8):1241-4. Japanese. PMID 8031168
- [Background] Surawicz CM, Elmer GW, Speelman P, McFarland LV, Chinn J, van Belle G. Prevention of antibiotic-associated diarrhea by Saccharomyces boulardii: a prospective study. Gastroenterology. 1989 Apr;96(4):981-8. doi: 10.1016/0016-5085(89)91613-2. PMID 2494098
- [Background] Salek T, Mardiak J, Obertova J, Sycova-Mila Z, Koza I. New weekly schedule of irinotecan as second line treatment in advanced colorectal cancer. Proc Am Soc Clin Oncol 21: 2378, 2002.
- [Background] Talbot GH, Cassileth PA, Paradiso L, Correa-Coronas R, Bond L. Oral enoxacin for infection prevention in adults with acute nonlymphocytic leukemia. The Enoxacin Prophylaxis Study Group. Antimicrob Agents Chemother. 1993 Mar;37(3):474-82. doi: 10.1128/AAC.37.3.474. PMID 8460916
- [Background] Vandenplas Y. Bacteria and yeasts in the treatment of acute and chronic infectious diarrhea. Part I. Bacteria. Clin Microbiol Infect. 1999 Jun;5(6):299-307. doi: 10.1111/j.1469-0691.1999.tb00148.x. PMID 11856274
- [Background] Viaud S, Saccheri F, Mignot G, Yamazaki T, Daillere R, Hannani D, Enot DP, Pfirschke C, Engblom C, Pittet MJ, Schlitzer A, Ginhoux F, Apetoh L, Chachaty E, Woerther PL, Eberl G, Berard M, Ecobichon C, Clermont D, Bizet C, Gaboriau-Routhiau V, Cerf-Bensussan N, Opolon P, Yessaad N, Vivier E, Ryffel B, Elson CO, Dore J, Kroemer G, Lepage P, Boneca IG, Ghiringhelli F, Zitvogel L. The intestinal microbiota modulates the anticancer immune effects of cyclophosphamide. Science. 2013 Nov 22;342(6161):971-6. doi: 10.1126/science.1240537. PMID 24264990
- [Background] Wiernik PH, Banks PL, Case DC Jr, Arlin ZA, Periman PO, Todd MB, Ritch PS, Enck RE, Weitberg AB. Cytarabine plus idarubicin or daunorubicin as induction and consolidation therapy for previously untreated adult patients with acute myeloid leukemia. Blood. 1992 Jan 15;79(2):313-9. PMID 1730080
- [Background] Wunderlich PF, Braun L, Fumagalli I, D'Apuzzo V, Heim F, Karly M, Lodi R, Politta G, Vonbank F, Zeltner L. Double-blind report on the efficacy of lactic acid-producing Enterococcus SF68 in the prevention of antibiotic-associated diarrhoea and in the treatment of acute diarrhoea. J Int Med Res. 1989 Jul-Aug;17(4):333-8. doi: 10.1177/030006058901700405. PMID 2676650
- [Background] Bishop JF, Matthews JP, Young GA, Szer J, Gillett A, Joshua D, Bradstock K, Enno A, Wolf MM, Fox R, Cobcroft R, Herrmann R, Van Der Weyden M, Lowenthal RM, Page F, Garson OM, Juneja S. A randomized study of high-dose cytarabine in induction in acute myeloid leukemia. Blood. 1996 Mar 1;87(5):1710-7. PMID 8634416
- [Result] Allen SJ, Okoko B, Martinez E, Gregorio G, Dans LF. Probiotics for treating infectious diarrhoea. Cochrane Database Syst Rev. 2004;(2):CD003048. doi: 10.1002/14651858.CD003048.pub2. PMID 15106189